CLINICAL TRIAL: NCT07041177
Title: Evaluation of the Efficacy and Safety of NeoThelium FT Amnion Skin Graft in the Management of Chronic Open Wounds: A Prospective Case Series
Brief Title: Prospective Case Series Evaluating the Efficacy and Safety of NeoThelium FT for Open Wounds
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NuScience Medical Biologics, LLC (Industry)
Collaborators: SygNola, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NeOpen
Record Dates: First submitted 2025-06-19; First posted 2025-06-27 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Open Wound
Keywords: Chronic Wounds; Cellular, Acellular, Matrix-like Product (CAMP); Cellular and/or Tissue Product (CTP); Dehydrated Complete Human Placental Membrane (dCHPM)

STUDY DESIGN:
Intervention Model Description: NeoThelium FT in addition to Standard of Care
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NeoThelium FT + SOC (Experimental): Wound cleansing, sharps debridement, NeoThelium FT application, Dressing for moisture balance, Offloading
  Interventions: Other: NeoThelium FT

INTERVENTIONS:
Other: NeoThelium FT — NeoThelium FT is a dehydrated wound covering derived from donated human placental tissue. NeoThelium FT is a dual-layer membrane with amnion and chorion combination layers.

SUMMARY:
This is a prospective case series evaluating the efficacy and safety of NeoThelium FT Amnion Skin Graft in the Mangement of Open Wounds

DETAILED DESCRIPTION:
This research will take place across multiple medical centers, where both researchers and participants will know which treatment is being used (open label). Patients who agree to participate and meet the study requirements during screening will begin SOC plus NeoThelium FT weekly applications. The subject will continue follow-up per the original schedule. As this is a post-marketing study, it will gather information regarding the efficacy of treatment while also supporting insurance reimbursement decisions.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, 18 years of age or older
2. Subject has a medical diagnosis of "other" Open wound
3. Subject has a chronic open wound present for 4 weeks or greater (documented in medical record)
4. Ulcer area is a minimum of 1 cm2 and a maximum of 25 cm2 at first treatment visit
5. Index wound has a maximum depth of 1cm at the first treatment visit
6. Subject is able and willing to follow the protocol requirements
7. Subject had signed informed consent
8. Adequate circulation if wound is location on the lower extremity demonstrated by an ABI of >0.7 and <1.3, or TBI of >0.6 within 30 days prior to informed consent OR an arterial ultrasound noted with patent circulation and without significant stenosis 90 days prior to the first treatment visit.
9. The chronic open wound is treated with offloading therapy at the Principal Investigator's discretion, if applicable to location, while standing, sitting, and lying down for 7 days prior to the first treatment visit
10. Wound free of clinical infection or clinically visible exposed bone (no purulent discharge, cellulitis, or osteomyelitis) 7 days prior to treatment visit 1

Exclusion Criteria:

1. Subject is unable to comply with protocol treatment
2. Subject with a wound diagnosis of diabetic foot wound, pressure wound, venous leg wound, burn wound, or alternative diagnosis other than "open wound"
3. Presence of systemic infection, sepsis, or osteomyelitis at screening.
4. Multiple wounds at the same site of the referenced wound with < 2 cm separation from the target ulcer.
5. Subject has major uncontrolled medical disorders in the opinion of the investigator, such as serious cardiovascular, renal, liver, pulmonary, autoimmune, palliative care, or inherited blood disorders that may affect wound healing.
6. Subject actively being treated for malignant disease or history of malignancy or radiation therapy at the site of wound.
7. Subject has comorbid conditions that may compromise subject safety in the opinion of the investigator
8. Known contraindications or hypersensitivity to amniotic membrane products or components of NeoThelium FT.
9. Concurrent participation in alternative clinical trial that involves investigational drug or HCT/P interfering with wound treatment and/or healing.
10. Subject is pregnant or breastfeeding
11. Subject with history of immunosuppressant treatment (systemic corticosteroids >10mg daily dose), cytotoxic chemotherapy, or topical steroid application to the ulcer surface for >2 weeks duration within 30 days prior to the first treatment visit; or anticipated use of the above during the course of the study
12. Wound previously treated with CAMPs, tissue engineered, or scaffold materials within 30 days prior to enrollment
13. Index ulcer suspicious of neoplasm in the opinion of the principal investigator
14. Open wound with active infection
15. Wound depth with visible exposed bone
16. Index wound suspicious of neoplasm in the opinion of the principal investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08-25 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Complete Wound Closure | 1-14 weeks
  The primary endpoint will be the percentage of target ulcers that achieve complete wound closure.

SECONDARY OUTCOMES:
Percentage Wound Area Change | 1-12 weeks
  The percentage change in wound area from TV-1 to TV-13 will be measured weekly using standardized method of wound area measurement and physical examination.
Follow-Up Closure | 2 weeks
  Number of wounds remaining closed during the 2-week follow-up
Time to Closure | 1-12 weeks
  Average number of grafts/weeks used to achieve wound closure

CONTACTS AND LOCATIONS:
Overall Officials: Angelina Ferguson, DNP, Study Chair — SygNola, LLC
Locations (1):
- MedCentris of Hammond, Hammond, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No